CLINICAL TRIAL: NCT02463461
Title: Comparison Between Multiple Wrist-worn Actigraphy Devices and Polysomnography
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not sure if we are going to do this study now.
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Weill Cornell Medical College in Qatar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1406015180
Record Dates: First submitted 2015-01-13; First posted 2015-06-04 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- ActiSleep Activity Monitor (Experimental): Subjects placed in this group will given an ActiSleep Activity Monitor for the one night of the study.
  Interventions: Device: ActiSleep Activity Monitor
- Jawbone Activity Monitor (Experimental): Subjects placed in this group will given a Jawbone Activity Monitor for the one night of the study.
  Interventions: Device: Jawbone Activity Monitor
- Actiwatch 2 Activity Monitor (Experimental): Subjects placed in this group will given an Actiwatch 2 Activity Monitor for the one night of the study.
  Interventions: Device: Actiwatch 2 Activity Monitor
- FitBit Activity Monitor (Experimental): Subjects placed in this group will given a FitBit Activity Monitor for the one night of the study.
  Interventions: Device: FitBit Activity Monitor
- Actigraph by Ambulatory Monitoring Activity Monitor (Experimental): Subjects placed in this group will given an Actigraph by Ambulatory Monitoring Activity Monitor for the one night of the study.
  Interventions: Device: Actigraph by Ambulatory Monitoring Activity Monitor

INTERVENTIONS:
Device: ActiSleep Activity Monitor — Subjects in this group will wear a ActiSleep Activity Monitor.
  Arms: ActiSleep Activity Monitor
Device: Jawbone Activity Monitor — Subjects in this group will wear a Jawbone Activity Monitor.
  Arms: Jawbone Activity Monitor
Device: Actiwatch 2 Activity Monitor — Subjects in this group will wear a Actiwatch 2 Activity Monitor.
  Arms: Actiwatch 2 Activity Monitor
Device: FitBit Activity Monitor — Subjects in this group will wear a FitBit Activity Monitor.
  Arms: FitBit Activity Monitor
Device: Actigraph by Ambulatory Monitoring Activity Monitor — Subjects in this group will wear a Actigraph by Ambulatory Monitoring Activity Monitor.
  Arms: Actigraph by Ambulatory Monitoring Activity Monitor

SUMMARY:
The primary objective of the proposed study is to investigate the agreement levels of modern and well-established actigraphy devices against PSG in healthy as well as patient populations for multiple sleep parameters across two study sites (Qatar and New York City).

DETAILED DESCRIPTION:
The importance of sleep upon physiological and psychological health has been extensively documented. It has been proposed that adequate sleep, as well as good sleep quality, is vital for wellbeing. (1). Some have suggested that sleep curtailment has paralleled the increased prevalence of cardiometabolic disease including obesity (2), type 2 diabetes mellitus (3, 4), hypertension (5, 6) and more. Sleep researchers face a major challenge since there are multiple methods for sleep assessment, all of which have advantages and disadvantages.Whilst polysomnography (PSG) is considered to be the gold standard for sleep assessment, there are some limitations including laboratory attendance for the participant and sleep scoring variance. Sleep questionnaires are widely utilized, particularly in large epidemiological studies, but are susceptible to inaccuracies and some have not been validated against PSG. Wrist actigraphy has provided researchers with an attractive equivalent and there are now multiple commercial manufacturers available. Actigraphic devices are usually worn on the non-dominant wrist and the instrument is used to monitor wrist movements through the use of an accelerometer and a memory chip. Wrist actigraphy is useful in the detection of sleep, wake, and activity.

ELIGIBILITY:
Inclusion Criteria:

* Attending a regularly scheduled Polysomnography test at Weill Cornell Medical College. Male or female. 18-80 years old

Exclusion Criteria:

* Not attending a regularly scheduled Polysomnography test at Weill Cornell Medical College. Under 18 or over 80 years old. Pregnancy. Unable to provide informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-08; Primary Completion 2017-07 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Total sleep time (TST) | 1 night
  The amount of actually sleep time in a sleep episode; this time is equal to the total sleep episode less the awake time. TST is the total of all REM and NREM sleep in a sleep episode.

SECONDARY OUTCOMES:
Wake After Sleep Onset (WASO) | 1 Year
  (Wake After Sleep Onset) Total minutes of wakefulness recorded after Sleep Onset, as scored by epochs.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Krieger, Principal Investigator — Weill Medical College of Cornell University

IPD SHARING:
Plan to Share IPD: Undecided